CLINICAL TRIAL: NCT05577117
Title: Opioid Free Anesthesia Versus Opioid Based Anesthesia for Improvement of the Surgical Field Condition in Elderly Patients Undergoing Arthroscopic Shoulder Surgery. A Randomized Comparative Study
Brief Title: Fentanyl vs Dexmedetomidine for Arthriscopic Shoulder Intervention in Elderly.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Ismail, Lecturer of Anesthesia, Surgical ICU and pain management at Faculty of medicine Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MS-201-2022
Record Dates: First submitted 2022-09-26; First posted 2022-10-13 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Lesions
MeSH Terms: interventions — Dexmedetomidine; Acetaminophen; Fentanyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid free (OFA) group (Active Comparator): 1000 mg paracetamol + dexmedetomidine 1 µg/kg over 10 min as loading dose and dexamethasone 0.1 mg/kg and lidocaine 1 mg/kg IV bolus Then continuous infusion of dexmedetomidine at a rate of 0.5 µg/kg/h with lidocaine 2 mg/kg/hr and magnesium sulfate 1.5 g/hr during surgery .
  Interventions: Drug: Dexmedetomidine
- fentanyl (F) group (No Intervention): fentanyl 2 µg/kg as loading dose followed by continuous infusion at a rate of 1 µg/kg/h during surgery.

INTERVENTIONS:
Drug: Dexmedetomidine — drugs are injected with induction of general anesthesia
  Other Names: paracetamol; fentanyl
  Arms: opioid free (OFA) group

SUMMARY:
Arthroscopic shoulder surgeries are commonly used as a minimally invasive surgery for shoulder diseases. however, it causes moderate-to-severe pain and needs stabilization of hemodynamics, without compromising the patient, to the degree that lessens the intraarticular bleeding to provide adequate visualization by the surgeon owing to inability to use a tourniquet in this situation.

Opioids have known side effects, like respiratory depression, postoperative nausea and vomiting, pruritus, difficulty in voiding, and ileus. These complications may lead to a prolonged hospital stay.

The elderly patients are predisposed to a greater hemodynamic changes due to the higher resting sympathetic tone ,altered beta receptor sensitivity , depleted intravascular volume because of frequent use of diuretics, increased myocardial stiffness ,increased arterial stiffness, reduced sinus node function and baroreceptor responsiveness and other patients comorbidities. So they are at increased risk complications as myocardial infarction, stroke and delirium.

Opioid free anesthesia is a technique with no opioids administered intraoperatively through either systemic, neuraxial, or tissue infiltration routes. The number of case reports and small prospective studies from all over the world supports its benefits.

OFA depends on combinations of non-opioid agents and adjuncts, including lidocaine, magnesium, dexmedetomidine, ketamine,and dexamethasone to produce anesthesia, and analgesia.

Dexmedetomidine is an a2 agonist that possesses anxiolytic, anesthetic, hypnotic, and analgesic properties. In addition, it reduces the pressor responses mediated by the sympathetic nervous system.

Lignocaine is a short-acting amide local anaesthetic agent. It is potent as a sodium channel blocker and has been shown to provide excellent analgesia when administered intravenously . The evidence base supports lignocaine as an analgesic agent, an opioid-sparing agent, an anti-inflammatory and a co-anaesthetic.

n,Complex regional pain syndrome,opioid-tolerant patient and early recovery after surgery, however, few studies focused on its ablility to improve the surgical field condition which depends on the hemodynamics especially in elderly patients.

Aim is to Compare OFA with Opioid anesthesia (OA) as regards improvement of the surgical field condition in elderly patients undergoing arthroscopic shoulder surgery under general anesthesia.

DETAILED DESCRIPTION:
Arthroscopic shoulder surgeries are commonly used as a minimally invasive surgery for shoulder diseases. however, it causes moderate-to-severe pain and needs stabilization of hemodynamics, without compromising the patient, to the degree that lessens the intraarticular bleeding to provide adequate visualization by the surgeon owing to inability to use a tourniquet in this situation.

Controlling the pain in shoulder surgery facilitates early mobilization, fast functional recovery and allows pain-free muscle contraction.

Opioids have known side effects, like respiratory depression, postoperative nausea and vomiting, pruritus, difficulty in voiding, and ileus. These complications may lead to a prolonged hospital stay.

The elderly patients are predisposed to a greater hemodynamic changes due to the higher resting sympathetic tone ,altered beta receptor sensitivity , depleted intravascular volume because of frequent use of diuretics, increased myocardial stiffness ,increased arterial stiffness, reduced sinus node function and baroreceptor responsiveness and other patients comorbidities. So they are at increased risk complications as myocardial infarction, stroke and delirium.

Opioid free anesthesia is a technique with no opioids administered intraoperatively through either systemic, neuraxial, or tissue infiltration routes. The number of case reports and small prospective studies from all over the world supports its benefits.

Initially, OFA depends on combinations of non-opioid agents and adjuncts, including lidocaine, magnesium, dexmedetomidine, ketamine,and dexamethasone to produce anesthesia, and analgesia.

Magnesium is a non-competitive antagonist of N-methyl-D-aspartate (NMDA) and has anti-inflammatory effects because it decreases interleukin 6 (IL-6) and tumour necrosis factor (TNF-alpha) levels postoperatively.

Dexamethasone is a mineraloglucocorticoid that has been shown to be effective as an antiemetic in a number of surgical operations. Dexamethasone was integrated into the multimodal opioid-free approach based on De Oliveira's and others' findings that dosages of> 0.1 mg/kg exhibit clinically significant analgesic characteristics in lean adults.

Ketamine is another non-competitive antagonist of the n-methyl-D-aspartate receptor and is commonly used either as a small bolus of 0.25-0.5 mg/kg IBW or in a low-dose continuous infusion at 2-2.5 μg/kg/min. Schug and others have summarised its benefits in APMSE4 in both the general acute pain population and bariatric patients.

Dexmedetomidine is an a2 agonist that possesses anxiolytic, anesthetic, hypnotic, and analgesic properties. In addition, it reduces the pressor responses mediated by the sympathetic nervous system.

Lignocaine is a short-acting amide local anaesthetic agent. It is potent as a sodium channel blocker and has been shown to provide excellent analgesia when administered intravenously . The evidence base supports lignocaine as an analgesic agent, an opioid-sparing agent, an anti-inflammatory and a co-anaesthetic.

n ,Complex regional pain syndrome ,opioid-tolerant patient and early recovery after surgery , however, few studies focused on its ability to improve the surgical field condition which depends on the hemodynamics especially in elderly patients.

Aim of the work is to Compare OFA with Opioid anesthesia (OA) as regards improvement of the surgical field condition in elderly patients undergoing arthroscopic shoulder surgery under general anesthesia.

Hypothesis :

The hemodynamics of the opioid free regimen will provide a better surgical field condition.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* aged > 65 years
* undergoing arthroscopic shoulder surgery under general anesthesia.

Exclusion Criteria:

* uncontrolled systemic diseases
* significant organ dysfunctions
* morbid obesity (BMI >35)
* history of allergy to the study drugs
* use of beta blockers
* chronic use of opioids

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
change in MBP | at start of the study drug infusion (Time1), after intubation (Time2), then every 10 min till the end of surgery. In the PACU will be recorded on arrival, after 30 min, 1 hour, and 2 hours.
  measuring mean blood pressure

SECONDARY OUTCOMES:
change in SBP | at start of the study drug infusion (Time1), after intubation (Time2), then every 10 min till the end of surgery. In the PACU will be recorded on arrival, after 30 min, 1 hour, and 2 hours.
  measuring systolic blood pressure
change in HR | at start of the study drug infusion (Time1), after intubation (Time2), then every 10 min till the end of surgery. In the PACU will be recorded on arrival, after 30 min, 1 hour, and 2 hours.
  measuring heart rate
Grades of surgical field bleeding, correlation between the difference in MAP and the grade of the surgical field. | 1 minute after visualizing the field with the arthroscope and then every 10 min till the end of surgery
  Grades of surgical field bleeding, correlation between the difference in MAP and the grade of the surgical field.
AMT score | after recovery from anesthesia (PACU AMT), 6 hours after surgery (Day-0) and on the next three postoperative days (Day-1, Day-2 and Day-3) at the same time of evaluation on day 0.
  AMT score
Postoperative complications as nausea, vomiting, bradycardia, hypoxia, shivering and delirium | within 2 hours in the PACU
  Postoperative complications as nausea, vomiting, bradycardia, hypoxia, shivering and delirium

CONTACTS AND LOCATIONS:
Overall Officials: Dalia K Ismail, Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol is shared and results and discussions will be shared once statistical analysis is done
Supporting Information: Study Protocol, CSR
Time Frame: Data should be available within 1 to 2 months
Access Criteria: Open